CLINICAL TRIAL: NCT00772018
Title: A Qualitative Study of Patients With Non-Invasive Bladder Cancer
Brief Title: Quality of Life and Symptom Management in Patients With Bladder Cancer
Status: Completed | Type: Observational
Sponsor: David Latini (Other)
Responsible Party: Sponsor-Investigator, David Latini, Assistant Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Other Study IDs: CDR0000600591; BCM-H-21570
Record Dates: First submitted 2008-10-12; First posted 2008-10-15 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Learning about quality of life and symptom management in patients with bladder cancer may help doctors learn about the effects of treatment and plan the best treatment.

PURPOSE: This clinical trial is studying of quality of life and symptom management in patients with bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To identify aspects of health-related quality of life (HRQOL) and symptom management in patients with non-invasive, low- or high-risk bladder cancer.
* To obtain feedback on data collection methods to enhance acceptability in these patients.

OUTLINE: Patients undergo a 10-minute screening in person or by phone to obtain demographic data and medical information (e.g., bladder cancer diagnosis and treatment history). Additional information is obtained from the clinical databases at the Baylor College of Medicine and the Michael E. DeBakey Veterans Affairs Medical Center. Patients who are eligible for the study are added to a waiting list for 1 of 4 focus groups based on disease status (high-risk or low-risk non-invasive bladder cancer) and gender. Patients participate in a 1.5- to 2-hour focus group discussion about the impact of bladder cancer on their quality of life and relationships. Patients receive information about community and Internet-based resources at the end of each group session.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of bladder cancer within the past 4 years

  * Non-invasive disease
  * Low- or high-risk disease
* Recruited from patients at the Baylor College of Medicine Scott Department of Urology clinics, the Michael E. DeBakey Veteran Affairs Medical Center, and the Urology Clinic at MD Anderson Cancer Center OR from participants at a community event

PATIENT CHARACTERISTICS:

* Not pregnant
* Able to read, speak, and understand English

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urology specialty clinic
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2008-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (HRQOL) and symptom management in patients with bladder cancer | One timepoint
  Study is a retrospective qualitative study of nonmuscle-invasive bladder cancer patients using a semi-structured interview protocol.

CONTACTS AND LOCATIONS:
Overall Officials: David M. Latini, PhD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Dan L. Duncan Cancer Center at Baylor College of Medicine, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas